CLINICAL TRIAL: NCT04829149
Title: A Cohort Study for Comparison of Statin Monotherapy and Rosuzet Tab.(Rosuvastatin/Ezetimibe) Administration and Statin Prescription Patterns in Patients With Dyslipidemia in Korea.
Brief Title: Statin Monotherapy and Rosuzet Tab.(Rosuvastatin/Ezetimibe) Administration in Patients With Dyslipidemia in Korea
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-ROZ-OS-01
Record Dates: First submitted 2021-03-22; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Dyslipidemias
Keywords: Statin; Rosuvastatin; New onset DM; LDL-C
MeSH Terms: conditions — Dyslipidemias | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Statin therapy group (No interventional): Observational. Statin therapy group: Once daily administered per the locally approved product information of rosuvastatin, simvastatin, atorvastatin, pitavastatin etc,. (except Rosuzet Tab.)
  Interventions: Other: Observational
- Rosuzet tablet group (No interventional): Observational. Rosuzet Tab.(ezetimibe/rosuvastatin) group: once daily administered per the locally approved product information of Rosuzet Tab. 10/5mg, 10/10mg, 10/20mg
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Statin therapy group and Rosuzet tablet group

SUMMARY:
A Cohort Study for Comparison of Statin Monotherapy and Rosuzet Tab.(Rosuvastatin/Ezetimibe) Administration and Statin Prescription Patterns in Patients With Dyslipidemia in Korea.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the effect of reducing LDL-C levels after 12 months of administration of Statin Monotherapy or Rosuzet Tab.(Rosuvastatin/Ezetimibe) in patients with dyslipidemia in Korea

ELIGIBILITY:
Inclusion Criteria:

1. Age≥19
2. Subject who is taking or is scheduled to take Statins therapy or Rosuzet Tab.
3. Not diagnosed with diabetes
4. Subject who can written informed consent voluntarily
5. Subject can continue to participate for 12 months on Study

Exclusion Criteria:

1. Patients for whom use of Rosuzet Tab. and Statin therapy is prohibited (e.g. patient who are hypersensitive to the main or compositional component of this drug, patient with active liver disease, patient with severe renal failure, patient using combinations with cyclosporin)
2. A pregnant or nursing woman

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A Korean dyslipidemia patient who is taking or is scheduled to take statins therapy or Rosuzet tablets
Sampling Method: Non-Probability Sample
Enrollment: 5717 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Lipid profiles | 12 months
  LDL-C percentage of change in Statin therapy group and Rosuzet group from baseline

SECONDARY OUTCOMES:
Lipid profiles | 6 months
  LDL-C percentage of change in Statin therapy group and Rosuzet group from baseline
Lipid profiles | 6, 12 months
  Triglyceride, HDL-C, Total Cholesterol percentage of change in Statin therapy group and Rosuzet group from baseline
Occurrence and aspect of new onset diabetes and adverse events | 12 months
  Occurrence and aspect of new onset diabetes and adverse events in Statin therapy group and Rosuzet group during the study period
Prescription rate | 12 months
  Prescription rate of Statin therapy group and Rosuzet group during the study period
Reason for medication change | 12 months
  Evaluation of Rate on reason for medication change in Statin therapy group and Rosuzet group during the study period
Medication compliance | 12 months
  MPR(medication possession ratio) of Statin therapy group and Rosuzet group during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Jeung KIM, Study Director — Hanmi Pharmaceutical Company Limited
Locations (1):
- Hanmi Pharmaceutical Company Limited, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No